CLINICAL TRIAL: NCT02141763
Title: A Subject-blind, Investigator-blind, Randomized, Placebo-controlled Study Evaluating the Safety, Pharmacokinetics, and Pharmacodynamics of Multiple Doses of UCB4940 in Subjects With Psoriatic Arthritis
Brief Title: Multiple Dose Study of UCB4940 in Subjects With Psoriatic Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Celltech (Industry)
Collaborators: Parexel (Industry); MAC Clinical Research (Other); Comac Medical (Industry); ARENSIA, Moldova (Unknown)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PA0007; 2013-004949-16 (EudraCT Number)
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — bimekizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 240/160/160 mg of UCB4940 (Experimental): 240 mg loading dose + 160 mg maintenance dose every 3 weeks on 2 occasions (total 3 doses)
  Interventions: Drug: UCB4940 160 mg; Drug: UCB4940 240 mg; Other: Placebo
- 160/80/80 mg of UCB4940 (Experimental): 160 mg loading dose + 80 mg maintenance dose every 3 weeks on 2 occasions (total 3 doses)
  Interventions: Drug: UCB4940 80 mg; Drug: UCB4940 160 mg; Other: Placebo
- 80/40/40 mg of UCB4940 (Experimental): 80 mg loading dose + 40 mg maintenance dose every 3 weeks on 2 occasions (total 3 doses)
  Interventions: Drug: UCB4940 40 mg; Drug: UCB4940 80 mg; Other: Placebo
- 560/320/320 mg of UCB4940 (Experimental): 560 mg loading dose + 320 mg maintenance dose every 3 weeks on 2 occasions (total 3 doses)
  Interventions: Drug: UCB4940 320 mg; Drug: UCB4940 560 mg; Other: Placebo
- Placebo (Placebo Comparator): 0.9% sodium chloride aqueous solution (physiological saline, preservative free) of pharmacopoeia (USP/Ph.Eur) quality in a 10 mL glass vial
  Interventions: Drug: UCB4940 40 mg; Drug: UCB4940 80 mg; Drug: UCB4940 160 mg; Drug: UCB4940 240 mg; Drug: UCB4940 320 mg; Drug: UCB4940 560 mg

INTERVENTIONS:
Drug: UCB4940 40 mg — * Active Substance: UCB4940
  * Pharmaceutical Form: solution
  * Concentration: vials at 80 mg/mL will be diluted with 0.9 % sodium chloride to a final concentration calculated to achieve the correct dose
  * Route of Administration: intravenous
  Arms: 80/40/40 mg of UCB4940; Placebo
Drug: UCB4940 80 mg — * Active Substance: UCB4940
  * Pharmaceutical Form: solution
  * Concentration: vials at 80 mg/mL will be diluted with 0.9 % sodium chloride to a final concentration calculated to achieve the correct dose
  * Route of Administration: intravenous
  Arms: 160/80/80 mg of UCB4940; 80/40/40 mg of UCB4940; Placebo
Drug: UCB4940 160 mg — * Active Substance: UCB4940
  * Pharmaceutical Form: solution
  * Concentration: vials at 80 mg/mL will be diluted with 0.9 % sodium chloride to a final concentration calculated to achieve the correct dose
  * Route of Administration: intravenous
  Arms: 160/80/80 mg of UCB4940; 240/160/160 mg of UCB4940; Placebo
Drug: UCB4940 240 mg — * Active Substance: UCB4940
  * Pharmaceutical Form: solution
  * Concentration: vials at 80 mg/mL will be diluted with 0.9 % sodium chloride to a final concentration calculated to achieve the correct dose
  * Route of Administration: intravenous
  Arms: 240/160/160 mg of UCB4940; Placebo
Drug: UCB4940 320 mg — * Active Substance: UCB4940
  * Pharmaceutical Form: solution
  * Concentration: vials at 80 mg/mL will be diluted with 0.9 % sodium chloride to a final concentration calculated to achieve the correct dose
  * Route of Administration: intravenous
  Arms: 560/320/320 mg of UCB4940; Placebo
Drug: UCB4940 560 mg — * Active Substance: UCB4940
  * Pharmaceutical Form: solution
  * Concentration: vials at 80 mg/mL will be diluted with 0.9 % sodium chloride to a final concentration calculated to achieve the correct dose
  * Route of Administration: intravenous
  Arms: 560/320/320 mg of UCB4940; Placebo
Other: Placebo — * Pharmaceutical Form: solution
  * Concentration: 0.9 % sodium chloride
  * Route of Administration: intravenous
  Arms: 160/80/80 mg of UCB4940; 240/160/160 mg of UCB4940; 560/320/320 mg of UCB4940; 80/40/40 mg of UCB4940

SUMMARY:
A study of UCB4940 in subjects with psoriatic arthritis to evaluate the safety and body distribution of UCB4940 in those patients. Neither the patient nor the doctor will know the treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of adult-onset psoriatic arthritis made at least 6 months prior to Screening as defined by the Classification Criteria for Psoriatic Arthritis
* Subject must have active psoriatic lesions or a history of psoriatic skin lesions
* Subject must have active arthritis
* Subject has had inadequate response to at least 1 nonbiologic Disease-Modifying Antirheumatic Drug (DMARD) (which may include methotrexate [MTX]) and/or 1 approved biologic DMARD
* Subject must be taking concurrent MTX for at least 3 months at time of Screening, and be on a stable dose at least 4 weeks prior to Baseline
* Female subject must be postmenopausal (at least 1 year), permanently sterilized or, if of childbearing potential, must be willing to use at least 2 effective methods of contraception during the study period
* Subject has clinical laboratory test results within the reference ranges of the testing laboratory
* Subject has Electrocardiogram (ECG) values within the reference ranges of the testing laboratory

Exclusion Criteria:

* Subject has absolute neutrophil count <1.5×109/L, and/or lymphocyte count <1.0×109/L
* Subject has known viral hepatitis, has a positive test for hepatitis B surface antigen or is hepatitis C virus antibody positive
* Subject tests positive to human immunodeficiency virus (HIV)-1/2 antibody
* Subject has a past medical history or family history of primary immunodeficiency
* Subject is splenectomized
* Subject has had a severe infection requiring hospitalization and/or treatment with iv antibiotics in the 6 months before the Screening Visit
* Subject has a history of positive tuberculosis (TB) test or evidence of possible TB or latent TB infection at Screening
* Subject has a high risk of acquiring TB infection
* Subject has a history of alcoholism or drug/chemical abuse
* Subject has an active infection or has had a serious within 6 weeks before the first dose of Investigational Medicinal Product (IMP)
* Subject has renal or liver impairment at the Screening Visit
* Subject has active neoplastic disease or history of neoplastic disease within 5 years of study entry (except for basal or squamous cell carcinoma of the skin or carcinoma in situ which has been definitively treated with standard of care approaches and is considered cured at Screening)
* Subject has any other acute or chronic illness which, in the opinion of the Investigator or Study Physician, could pose a threat or harm to the subject
* Subjects must not have a diagnosis of any other inflammatory arthritis, eg, rheumatoid arthritis, sarcoidosis, or systemic lupus erythematosus
* Subject has a current or past history of gastrointestinal ulceration
* Subjects must not have a noninflammatory condition (eg, osteoarthritis or a known diagnosis of fibromyalgia) that in the Investigator's opinion is symptomatic enough to interfere with evaluation of the effect of IMP on the subject's primary diagnosis of Psoriatic Arthritis (PsA)
* Subject has received a live vaccination within 6 weeks before the Screening Visit or intends to have or will need a live vaccination during the course of the study or for the 3 months following last IMP dosing
* Subject has had an inadequate response to more than 1 approved biologic Drug-Modifying Antirheumatic Drug (DMARD)
* Subject has received any investigational drug or experimental procedure within 90 days or 5 half-lives whichever is the longer before the first dose of UCB4940

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration at steady state (CmaxSS) of UCB 4940 during the duration of the study (up to Day 141) | From Baseline to Day 141
  * Day 1: predose; 1 hour (hr), 1.5 hr, 5 hr, 12 hr, 24 hr postdose
  * Day 8, 15: 1 sample
  * Day 22: predose, 1 hr postdose
  * Day 43: predose; 1 hr, 1.5 hr, 5 hr, 12 hr, 24 hr postdose
  * Day 48, 57, 64, 85, 141: 1 sample
Minimum plasma concentration at steady state (CminSS) of UCB4940 during the duration of the study (up to Day 141) | From Baseline to Day 141
  * Day 1: predose; 1 hour (hr), 1.5 hr, 5 hr, 12 hr, 24 hr postdose
  * Day 8, 15: 1 sample
  * Day 22: predose, 1 hr postdose
  * Day 43: predose; 1 hr, 1.5 hr, 5 hr, 12 hr, 24 hr postdose
  * Day 48, 57, 64, 85, 141: 1 sample
Area under the curve at steady state (AUCtau) of UCB4940 during the duration of the study (up to Day 141) | From Baseline to Day 141
  * Day 1: predose; 1 hour (hr), 1.5 hr, 5 hr, 12 hr, 24 hr postdose
  * Day 8, 15: 1 sample
  * Day 22: predose, 1 hr postdose
  * Day 43: predose; 1 hr, 1.5 hr, 5 hr, 12 hr, 24 hr postdose
  * Day 48, 57, 64, 85, 141: 1 sample
Time to reach maximum plasma concentration at steady state (tmax) of UCB4940 during the duration of the study (up to Day 141) | From Baseline to Day 141
  * Day 1: predose; 1 hour (hr), 1.5 hr, 5 hr, 12 hr, 24 hr postdose
  * Day 8, 15: 1 sample
  * Day 22: predose, 1 hr postdose
  * Day 43: predose; 1 hr, 1.5 hr, 5 hr, 12 hr, 24 hr postdose
  * Day 48, 57, 64, 85, 141: 1 sample
Total Clearance (CL) of UCB4940 during the duration of the study (up to Day 141) | From Baseline to Day 141
  * Day 1: predose; 1 hour (hr), 1.5 hr, 5 hr, 12 hr, 24 hr postdose
  * Day 8, 15: 1 sample
  * Day 22: predose, 1 hr postdose
  * Day 43: predose; 1 hr, 1.5 hr, 5 hr, 12 hr, 24 hr postdose
  * Day 48, 57, 64, 85, 141: 1 sample
Volume of distribution (V) of UCB4940 during the duration of the study (up to Day 141) | From Baseline to Day 141
  * Day 1: predose; 1 hour (hr), 1.5 hr, 5 hr, 12 hr, 24 hr postdose
  * Day 8, 15: 1 sample
  * Day 22: predose, 1 hr postdose
  * Day 43: predose; 1 hr, 1.5 hr, 5 hr, 12 hr, 24 hr postdose
  * Day 48, 57, 64, 85, 141: 1 sample
Percentage of subjects with at least one Treatment Emergent Adverse Event (TEAE) during the study | From Baseline to Day 141

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (3):
- 001, Sofia, Bulgaria
- 002, Saint Chisinau, Moldova
- 003, Manchester, United Kingdom

REFERENCES:
- [Derived] Glatt S, Baeten D, Baker T, Griffiths M, Ionescu L, Lawson ADG, Maroof A, Oliver R, Popa S, Strimenopoulou F, Vajjah P, Watling MIL, Yeremenko N, Miossec P, Shaw S. Dual IL-17A and IL-17F neutralisation by bimekizumab in psoriatic arthritis: evidence from preclinical experiments and a randomised placebo-controlled clinical trial that IL-17F contributes to human chronic tissue inflammation. Ann Rheum Dis. 2018 Apr;77(4):523-532. doi: 10.1136/annrheumdis-2017-212127. Epub 2017 Dec 23. PMID 29275332